CLINICAL TRIAL: NCT01902537
Title: Health Related Quality of Life in Female Patients With Chronic Constipation
Brief Title: An Observational Study to Evaluate the Quality of Life in Korean Female Participants With Chronic Constipation
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100894; PRUCRC4001
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Constipation
Keywords: Constipation; Prucalopride
MeSH Terms: conditions — Constipation | interventions — prucalopride; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants With Constipation: Participants with constipation receiving prucalopride will be observed for for the health related quality of life (QoL).
  Interventions: Drug: Prucalopride; observational study

INTERVENTIONS:
Drug: Prucalopride; observational study — This is an observational study. Korean female participants with chronic constipation and having received treatment previously will be assessed for the health related QoL.

SUMMARY:
The purpose of this observational study is to investigate health related quality of life (QoL) in Korean female participants with chronic constipation (long term decreased number of or difficulty making bowel movements) having received treatment previously.

DETAILED DESCRIPTION:
This is a cross-sectional (studies in which the presence or absence of disease or other health-related variables are determined in each member of the study population or in a representative sample at 1 particular time) observational study (a scientific study to make a clear and easy understanding of the cause and effect relationship) to investigate the health related QoL in Korean female participants with chronic constipation having received treatment previously by using EQ-5D (EuroQol 5 Dimension), SF-36 (Short Form Health Survey) and PAC-QoL (Patient Assessment of Constipation) questionnaires. The duration of study will be 6 months. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

-Korean female participants with chronic constipation having received treatment previously

Exclusion Criteria:

* Male participants
* Participants with psychological disease (disorders of the mind, thoughts, and behavior)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean female participants with chronic constipation, having received treatment previously for constipation. Participants who have visited Constipation Clinic of AMC or Department of Gastrointestinal for constipation therapy will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
EQ-5D-3L (EuroQol 5 Dimension 3 Level) Quality of life (QoL) Score at Baseline | Baseline
  The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 3 levels; 1 indicates better health state (no problems); 3 indicate worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
EQ-5D-3L (EuroQol 5 Dimension) Quality of life (QoL) Score at Week 1 | Week 1
  The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 3 levels; 1 indicates better health state (no problems); 3 indicate worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
EQ-5D-5L (EuroQol 5 Dimension 5 Level) Quality of life (QoL) Score at Baseline | Baseline
  The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 5 levels (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and possible total score range -0.654 to 1.000; higher score indicates a better health state.
EQ-5D-5L (EuroQol 5 Dimension 5 Level) Quality of life (QoL) Score at Week 1 | Week 1
  The EQ-5D is a participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, using 5 levels (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and possible total score range -0.654 to 1.000; higher score indicates a better health state.
Short Form 36 (SF-36) Quality of life (QoL) Score | Baseline
  The SF-36 is a standardized survey evaluating 8 domains (consisting of 2 components; physical and mental) of functional health and well being: physical and social functioning, physical and emotional role (role-physical, role-emotional) limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Participant Assessment of Constipation Quality of Life (PAC-QoL) Scale Score | Baseline
  The PAC-QOL is composed of 28 items grouped into four subscales related to dissatisfaction (5 items), physical discomfort (4 items), psychosocial discomfort (8 items), and worries and concerns (11 items). Participants rated the severity of each symptom on a five-point scale from 0 (absent) to 4 (very severe), and scores are reported as an average total score or subscale score. The overall and all subscale scores range from 0 to 4, with lower scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Seoul, South Korea